CLINICAL TRIAL: NCT00999739
Title: A Sequential Vaccination Strategy With Conjugated and Polysaccharide Pneumococcal Vaccines Compared With Polysaccharide Vaccine in HIV- Infected Adults.
Brief Title: Conjugate And Polysaccharide Vaccines Compared With Polysaccharide Vaccine In Hiv-Infected Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Hospital Son Llatzer (Other); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Maria Penaranda, Hospital Son Dureta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Maria Penaranda
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-10

CONDITIONS: Pneumococcal Vaccines; HIV; HIV Infections
Keywords: pneumococcal vaccines; HIV; antibody response; antibody affinity; Antibody formation; Phagocytosis
MeSH Terms: conditions — HIV Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- two vaccines (Experimental): people allocated to arm two vaccines will receive one dose of heptavalent pneumococcal conjugate vaccine at day 0 and 23-valent polysaccharide vaccine at week4 , 110 HIV-infected people will be included Intervention: administration of two vaccines
  Interventions: Biological: Prevenar and Pneumo23
- One vaccine (Experimental): people allocated to arm one will receive only one doses of pneumococcal polysaccharide 23-valent vaccine. 110 HIV-infected adults will be included in this arm Intervention: administration of one vaccine
  Interventions: Biological: Prevenar and Pneumo23

INTERVENTIONS:
Biological: Prevenar and Pneumo23 — Two vaccines: participants will receive via intramuscular in deltoid one dose of conjugated heptavalent vaccine at day 0 (Prevenar, Wyeth-lederle)and one dose of 23valent polysaccharide vaccine (Pneumo23, AventisPasteur)at week4 One vaccine:participants will receive only one dose of 23valent polysaccharide vaccine at day 0.
  Other Names: Prevenar (heptavalent conjugated pneumococcal vaccine); Pneumo23 (23valent polysaccharide pneumococcal vaccine)

SUMMARY:
Randomised study comparing two pneumococcal vaccination strategies in HIV-infected adults with moderate immunossupression (CD4 between 200 and 500 cells/uL and viral load under 5logs), one with conjugated heptavalent vaccine(Prevenar, Wyeth-Lederle) followed by polysaccharide vaccine 4 weeks after (Aventis-Pasteur), and two with one dose of polysaccharide vaccine. Determination of secondary effects related to both vaccines and determination of antibody concentration (ELISA) and avidity (ELISA with thiocyanate) and opsonophagocytosis killing activity against the seven serotypes included in the heptavalent vaccine before vaccination, at 4 weeks, at 8 weeks, at48 weeks and 96 weeks. A sample of 220 HIV-infected adults (110 in each group) will be needed to detect differences of 10% for a type I error o 5% for a limited population of 2500 HIV-infected adults. The main hypothesis are :the immunogenicity of pneumococcal vaccination with conjugate and polysaccharide vaccines is superior to immunogenicity induced by polysaccharide vaccination alone(antibody concentration), the avidity and opsonophagocytosis induced by two vaccines is better than the one after polysaccharide vaccine alone, both vaccinations are safe.

DETAILED DESCRIPTION:
Randomised study comparing two pneumococcal vaccination strategies in HIV-infected adults with moderate immunossupression (CD4 between 200 and 500 cells/uL and viral load under 5logs), one with conjugated heptavalent vaccine(Prevenar, Wyeth-Lederle) followed by polysaccharide vaccine 4 weeks after (Aventis-Pasteur), and two with one dose of polysaccharide vaccine. A sample of 220 HIV-infected adults will be randomised to receive twe strategy one(110 patients) one dose of heptavalent conjugated vaccine at day 0 and one dose of polysaccharide vaccine at week 4 (in deltoid muscle); or strategy two (110 patients) one dose of polysaccharide vaccine at day 0. Secondary effects to the vaccines will be evaluated by phone interview 3 days after vaccinations.

Blood samples will be taken at day 0(before the first vaccine), at week 4 before the polysaccharide in the group one, and 4 weeks after the polysaccharide in the group two) and at week 8 in the group one, and at weeks 48 and 96 in both groups Antibody concentration , avidity, and opsonophagocytic killing activity will be measured in all the samples for serotypes 4,14,19F,23F,6B,18C,9V.

Antibody concentration , avidity, and opsonophagocytic killing activity will be compared between both vaccine groups, and between prevaccination and at 4,8, 48 and 96 weeks of vaccination. Risk factors associated to good antibody response (antibody duplication and antibody duplication plus achieve a level above 1ug/ml)will be measured at 8, 48 and96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adults with CD4 between 200 and 500 cels/ul and viral load under 5 logarithm

Exclusion Criteria:

* previous pneumococcal vaccine, pregnancy, advanced renal or liver disease, other vaccine or antibiotics 6 weeks before, other immunosuppression, immunoglobulins or investigation drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Antibody response in terms of antibody concentration at 4,8,48 and 69 weeks of vaccination | 4, 8, 48 and 96 weeks of vaccination

SECONDARY OUTCOMES:
Avidity of the antibodies induced in the two vaccination groups before and at 4 ,8 , 48 and 96 weeks of vaccination | 4 , 8 ,48 and 96 weeks after vaccintation
safety of both vaccines | 3 days
risk factors associated to a good vaccine response | 8 weeks, 48 weeks, 96 weeks
opsonophagocytic activity against the seven polysaccharides before, and after 4,8,48 and 96 weeks of vaccination | 4,8,48 and 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: maria penaranda, physician, Principal Investigator — Hospital Son Dureta; antonio payeras, physician, Principal Investigator — Hospital Son Llatzer
Locations (2):
- Spain (2):
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands

REFERENCES:
- [Derived] Penaranda M, Payeras A, Cambra A, Mila J, Riera M; Majorcan Pneumococcal Study Group. Conjugate and polysaccharide pneumococcal vaccines do not improve initial response of the polysaccharide vaccine in HIV-infected adults. AIDS. 2010 May 15;24(8):1226-8. doi: 10.1097/QAD.0b013e3283389de5. PMID 20299956